CLINICAL TRIAL: NCT06415214
Title: A Multicenter, Randomized, Double-blinded, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy and Safety of HRS-7535 in Adults With Diabetic Kidney Disease in Type 2 Diabetes
Brief Title: Efficacy and Safety of HRS-7535 Tablets in Adults With Diabetic Kidney Disease in Type 2 Diabetes
Acronym: SOLID-DKD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-7535-203
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-05

CONDITIONS: Diabetic Kidney Disease, Type 2 Diabetes
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A，Subjects will receive Placebo administered orally (Placebo Comparator)
  Interventions: Drug: Placebo
- Group B，Subjects will receive HRS-7535 administered orally (Experimental)
  Interventions: Drug: HRS-7535
- Group C，Subjects will receive escalated HRS-7535 administered orally (Experimental)
  Interventions: Drug: HRS-7535

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Group A，Subjects will receive Placebo administered orally
Drug: HRS-7535 — HRS-7535
  Arms: Group B，Subjects will receive HRS-7535 administered orally; Group C，Subjects will receive escalated HRS-7535 administered orally

SUMMARY:
The study is a 16-week multicenter, randomized, double-blind, placebo-controlled, parallel-designed Phase II clinical study. The aim of this trial is to evaluate the efficacy and safety of HRS-7535 in subjects with diabetic kidney disease in type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, 18-75 years of age at the time of signing informed consent;
2. Body weight ≥50 kg, 20.0 kg/m2 ≤BMI ≤40.0 kg/m2;
3. Diabetic kidney disease was diagnosed, and the eGFR≥30 mL/min/1.73 m2;
4. Had a history of T2DM at least 3 months, or had diabetic retinopathy as assessed by the investigators;
5. UACR ≥300 and <3000 mg/g;
6. HbA1c ≥6.5% and ≤10.0%;
7. ACEI/ARB was used for ≥3 months and ACEI/ARB was stabilized at either the maximum recommended dose (reference to the drug label) or the maximum tolerated dose within 4 weeks;
8. Use hypoglycemic drugs for ≥3 months (the dosage of SGLT2i remains stable if used);
9. Able and willing to provide a written informed consent;

Exclusion Criteria:

1. Have type 1 diabetes mellitus or specific type of diabetes;
2. Acute kidney injury or dialysis treatment within 6 months;
3. Kidney transplantation is planned during the trial;
4. History of acute cardiovascular and cerebrovascular diseases within 6 months prior to screening;
5. Any organ-system malignancies developed within 5 years except for cured local basal cell cancer of the skin and in-situ cancer of the cervix;
6. history of blood donation or blood loss in the 3 months before screening, or blood transfusion in the 2 months before screening;
7. Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using an adequate contraceptive method;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2024-06-21 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Ratio of UACR at week 16 to UACR at baseline | at Week 16

SECONDARY OUTCOMES:
24 hour urine analysis results at Week 16 | at Week 16
Proportion of subjects with a 30% decrease in UACR from baseline at Week 16 | at Week 16
Change from baseline in eGFR at Week 16 | at Week 16
Change from baseline in HbA1c at Week 16 | at Week 16
Proportion of subjects reaching the target of HbA1c (<7.0%、<6.5%) at Week 16 | at Week 16
Change from baseline in FPG at Week 16 | at Week 16
Change from baseline in insulin at Week 16 | at Week 16
Change from baseline in c-peptide at Week 16 | at Week 16
Change from baseline in body weight at Week 16 | at Week 16
Proportion of subjects receiving glycemic rescue medicine at Week 16 | at Week 16
A summary of adverse events, including serious adverse events (SAEs), and hypoglycemic event at Week 16 | at Week 16

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided